CLINICAL TRIAL: NCT05621278
Title: Children to Adults Mental and Psychosomatic Health Study (CAMPS): A Longitudinal Cohort Study
Brief Title: Children to Adults Mental and Psychosomatic Health Study (CAMPS)
Status: Recruiting | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, YinyinZang, Principal Investigator, Peking University
Other Study IDs: CAMPS
Record Dates: First submitted 2022-09-09; First posted 2022-11-18 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Mental Health Wellness; Cognitive Function; Physical Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Children: Grade 4 to 6 students (aged 9-12) in primary school.
- Adolescent: Grade 7 to 12 students (aged 12-18) in middle school and high school.
- Students' teachers: School Teachers
- Students' parents: Parents of students mentioned above.

SUMMARY:
This study titled the Children to Adults Mental and Psychosomatic Health Study (CAMPS), aims to explore the interplay between mental health, psychosomatic factors, and adverse childhood experiences (ACE) across a broad age range, from school-age children to adults in China. The study will involve participants from various educational settings, including teachers, students, and parents, who will be recruited through schools. The assessment methodology will combine validated psychometric scales and behavioral experiments to comprehensively evaluate mental and physical health aspects and the impact of ACEs. This integrative approach is designed to illuminate the complex relationships between psychological well-being, somatic symptoms, and early life stressors across different life stages.

ELIGIBILITY:
Inclusion Criteria:

1. Students from 5 grade to 12 grade, their parents and teachers
2. able to read, answer questionnaires and complete experiments.

Exclusion Criteria:

a. Students who suspend schooling.

Ages: 9 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Students from 5 grade to 12 grade and their parents and teachers in Chinese schools.
Sampling Method: Non-Probability Sample
Enrollment: 400000 (Estimated)
Dates: Start 2022-09-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Irritability | 1 month
  A 17-item irritability measurement scale, the Peking irritability scale, measures impulsive emotions, thoughts, and behaviors on a 5-point Likert scale (score from 1 to 5, and total score varies from 17 to 85). A higher score represents higher irritability.
Alexithymia | 1 month
  A 36-item Peking alexithymia scale measures thoughts and behaviors that prevent people from feeling or recognizing negative emotions on a 5-point Likert scale (1 to 5, and total scores vary from 36 to 180). A higher score represents more severe alexithymia.
Depression for adults | 2 weeks
  The 9-item patient health questionnaire (PHQ-9) for adults (score from 0 to 3, and total score varies from 0 to 27). A higher score represents worse depression symptoms.
Depression | 2 weeks
  Children's depression inventory (CDI) for adolescents and children (score from 0 to 2, and total score vary from 0 to 54). A higher score represents worse depression symptoms.
Generalized anxiety disorder | 2 weeks
  The Generalized Anxiety Disorder-7 scale (GAD-7) for adults, adolescents, and children (scored from 0 to 3, and total score from 0 to 21). A higher score represents worse anxiety symptoms.
Anxiety and depression for adolescents and children | 2 weeks
  The Revised Child Anxiety and Depression Scale (RCADS) for adolescents and children (scored from 0 to 3, and total score from 0 to 75). A higher score represents worse anxiety and depression symptoms.
PTSD for adults | 1 month
  The PTSD Symptoms Scale-Interview for DSM-5 (PSSI-5) for adults (score from 0 to 4, and total scores vary from 0 to 80). A higher score represents worse PTSD symptoms.
PTSD for adolescents and children | 1 month
  The Child PTSD Symptom Scale for DSM-5 (CPSS-5) for adolescents and children (scores from 0 to 4, and total scores vary from 0 to 80). A higher score represents worse PTSD symptoms.
NSSI | 1 year
  The non-suicidal self-injury assessment tool (NSSI-AT-Severity) for adolescents and children (total scores vary from 5 to 16). A higher score represents a worse self-injury situation.
Suicide | 1 year
  The suicidal behaviors questionnaire-revised (SBQ-R) for adolescents and children (total scores vary from 3 to 18). A higher score represents a higher suicide risk.
Emotion recognition | Half year
  The Morph task for adolescents to examine the emotion recognition capability.
Excutive function | Half year
  The Go/Nogo task for adolescents is to examine inhibition function.
Adverse Childhood Experiences (ACE) | each year
  A questionnaire measuring adverse childhood experiences with 26 items.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided